CLINICAL TRIAL: NCT02383745
Title: Integrating EEG Into Acute Medicine: EEG in In-hospital Patients With Seizure or Altered Mental State Who Have Been Consulted by Medical Emergency Team
Brief Title: EEG in In-hospital Patients With Seizure or Altered Mental State
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KUH507T011
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Status Epilepticus; Seizure; Altered Mental Status
Keywords: Acute EEG; status epilepticus; seizure
MeSH Terms: conditions — Status Epilepticus; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Acute EEG with fast EEG electrode

SUMMARY:
In Kuopio University Department of Clinical Neurophysiology there have been designed a fast EEG electrode, that is suitable for acute emergency use. It is easy to set up, records high quality EEG and can detect the most important EEG abnormalities comparable to conventional EEG. This study will address the clinical use of acute EEG with fast electrode set in in-hospital patients who have been consulted by Medical Emergency Team because of seizure or altered mental state of uncertain etiology. Patients are going to be treated in ICU and EEG monitoring will continue for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* In-hospital patients who have a seizure or altered mental state and are going to be treated in ICU

Exclusion Criteria:

* Patiets that are not going to be treated in ICU
* Patients with a Do Not Attempt to Resuscitate - decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In-hospital patients, who have seizure or altered mental state and have been consulted by MET-team
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Quantity of EEG abnormalities detected | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Esa Mervaala, MD, PhD,professor, Study Director — Professor in Clinical Neurophysiology
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland